CLINICAL TRIAL: NCT02329327
Title: Prospective, Open-Label Study of Andexanet Alfa in Patients Receiving a Factor Xa Inhibitor Who Have Acute Major Bleeding (ANNEXA-4)
Brief Title: A Study in Participants With Acute Major Bleeding to Evaluate the Ability of Andexanet Alfa to Reverse the Anticoagulation Effect of Direct and Indirect Oral Anticoagulants (Extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Portola Pharmaceuticals, LLC (a wholly owned subsidiary of Alexion Pharmaceuticals) (Industry); Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-505
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Bleeding
Keywords: Factor Xa Inhibitors; Major; Bleeding; Anticoagulant; Major Bleeding; Andexanet Alfa; Reversal Agent
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Andexanet (Experimental): Participants received andexanet as an intravenous bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
  Interventions: Biological: Andexanet

INTERVENTIONS:
Biological: Andexanet — There were 2 possible dosing regimens: Low dose = 400 milligram (mg) bolus plus 4 mg/minute continuous infusion for 120 minutes; High dose = 800 mg bolus plus 8 mg/minute continuous infusion for 120 minutes.
  Other Names: ALXN2070; Andexanet Alfa; PRT064445; Andexxa

SUMMARY:
The purpose of this study was to evaluate the hemostatic efficacy of andexanet alfa (andexanet) in participants receiving a factor Xa (FXa) inhibitor (apixaban, rivaroxaban, edoxaban, enoxaparin) who were experiencing an acute major bleed. The safety of andexanet was also studied.

ELIGIBILITY:
Key Inclusion Criteria:

1. Acute major bleeding episode that required urgent reversal of anticoagulation; defined by at least one of the following:

   * Acute bleeding that was potentially life-threatening, or
   * Acute bleeding associated with a fall in hemoglobin level by ≥2 grams/deciliter (g/dL), or
   * Acute bleeding associated with a hemoglobin level of ≤8 g/dL if no baseline hemoglobin was available, or
   * Acute bleeding in a critical area or organ such as intraspinal, pericardial, or intracranial.
2. If bleeding was intracranial or intraspinal, the participant must have undergone a head computed tomography (CT) or magnetic resonance imaging (MRI) scan demonstrating the bleeding.
3. Participant received or was believed to have received one of the following within 18 hours prior to andexanet administration: apixaban, rivaroxaban, edoxaban, or enoxaparin.
4. For participants with intracranial bleeding, there must be a reasonable expectation that andexanet treatment will commence within 2 hours of the baseline imaging evaluation.

Key Exclusion Criteria:

1. The participant was scheduled to undergo surgery in less than 12 hours, with the exception of minimally invasive surgery/procedures.
2. Participant with an intracerebral hemorrhage that had any of the following:

   * Glasgow coma score <7, or
   * Intracerebral hematoma >60 cubic centimeters as assessed by CT or MRI
3. Participants with visible, musculoskeletal or intra-articular bleeding as their qualifying bleed.
4. Expected survival of less than 1 month.
5. Recent history (within 2 weeks) of a diagnosed thrombotic event as follows: venous thromboembolism, myocardial infarction, disseminated intravascular coagulation, cerebral vascular accident, transient ischemic attack, unstable angina pectoris hospitalization or severe peripheral vascular disease within 2 weeks prior to Screening.
6. Severe sepsis or septic shock at the time of Screening.
7. Pregnant or a lactating female.
8. Participant received any of the following drugs or blood products within 7 days of Screening:

   * Vitamin K antagonist
   * Dabigatran
   * Prothrombin Complex Concentrate (PCC) products or recombinant factor VIIa (rfVIIa)
   * Whole blood, plasma fractions
9. Treated with an investigational drug <30 days prior to Screening.
10. Planned administration of PCC, fresh frozen plasma or rfVIIa from Screening until within 12 hours after the end of the andexanet infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (87):
- United States (23):
  - Clinical Study Site, Long Beach, California
  - Clinical Study Site, Los Angeles, California
  - Clinical Study Site, Orange, California
  - Clinical Study Site, Fort Lauderdale, Florida
  - Clinical Study Site, Jacksonville, Florida
  - Clinical Study Site, Sarasota, Florida
  - Clinical Study Site, Tampa, Florida
  - Clinical Study Site, Annapolis, Maryland
  - Clinical Study Site, Boston, Massachusetts
  - Clinical Study Site, Detroit, Michigan
  - Clinical Study Site, Royal Oak, Michigan
  - Clinical Study Site, Troy, Michigan
  - Clinical Study Site, St Louis, Missouri
  - Clinical Study Site, Rochester, New York
  - Clinical Study Site, Asheville, North Carolina
  - Clinical Study Site, Chapel Hill, North Carolina
  - Clinical Study Site, Raleigh, North Carolina
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Cleveland, Ohio
  - Clinical Study Site, Pittsburgh, Pennsylvania
  - Clinical Study Site, Austin, Texas
  - Clinical Study Site, Fort Worth, Texas
  - Clinical Study Site, Huntington, West Virginia
- Belgium (3):
  - Clinical Study Site, Brussels
  - Clinical Study Site, Genk
  - Clinical Study Site, Leuven
- Canada (2):
  - Clinical Study Site, Hamilton, Ontario
  - Clinical Study Site, Montreal, Quebec
- France (5):
  - Clinical Study Site, Clermont-Ferrand
  - Clinical Study Site, Grenoble
  - Clinical Study Site, Limoges
  - Clinical Study Site, Lyon
  - Clinical Study Site, Poitiers
- Germany (33):
  - Clinical Study Site, Altenburg
  - Clinical Study Site, Augsburg
  - Clinical Study Site, Berlin
  - Clinical Study Site, Bremen
  - Clinical Study Site, Celle
  - Clinical Study Site, Chemnitz
  - Clinical Study Site, Coburg
  - Clinical Study Site, Detmold
  - Clinical Study Site, Dresden
  - Clinical Study Site, Essen
  - Clinical Study Site, Göttingen
  - Clinical Study Site, Greifswald
  - Clinical Study Site, Halle
  - Clinical Study Site, Hamburg
  - Clinical Study Site, Hanover
  - Clinical Study Site, Heidelberg
  - Clinical Study Site, Hessen
  - Clinical Study Site, Jena
  - Clinical Study Site, Konstanz
  - Clinical Study Site, Leipzig
  - Clinical Study Site, Ludwigshafen
  - Clinical Study Site, Lübeck
  - Clinical Study Site, Mainz
  - Clinical Study Site, Minden
  - Clinical Study Site, Munich
  - Clinical Study Site, Münster
  - Clinical Study Site, Osnabrück
  - Clinical Study Site, Regensburg
  - Clinical Study Site, Sande
  - Clinical Study Site, Trier
  - Clinical Study Site, Tübingen
  - Clinical Study Site, Ulm
  - Clinical Study Site, Würzburg
- Japan (14):
  - Clinical Study Site, Fukuoka
  - Clinical Study Site, Gunma
  - Clinical Study Site, Hiroshima
  - Clinical Study Site, Ibaraki
  - Clinical Study Site, Izumisano
  - Clinical Study Site, Kobe
  - Clinical Study Site, Kumamoto
  - Clinical Study Site, Nagoya
  - Clinical Study Site, Sendai
  - Clinical Study Site, Shiwa-gun
  - Clinical Study Site, Suita
  - Clinical Study Site, Tokyo
  - Clinical Study Site, Yamaguchi
  - Clinical Study Site, Yokosuka
- Clinical Study Site, Amsterdam, Netherlands
- Spain (3):
  - Clinical Study Site, Barcelona
  - Clinical Study Site, Cáceres
  - Clinical Study Site, Madrid
- United Kingdom (3):
  - Clinical Study Site, Cardiff
  - Clinical Study Site, London
  - Clinical Study Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Connolly SJ, Milling TJ Jr, Eikelboom JW, Gibson CM, Curnutte JT, Gold A, Bronson MD, Lu G, Conley PB, Verhamme P, Schmidt J, Middeldorp S, Cohen AT, Beyer-Westendorf J, Albaladejo P, Lopez-Sendon J, Goodman S, Leeds J, Wiens BL, Siegal DM, Zotova E, Meeks B, Nakamya J, Lim WT, Crowther M; ANNEXA-4 Investigators. Andexanet Alfa for Acute Major Bleeding Associated with Factor Xa Inhibitors. N Engl J Med. 2016 Sep 22;375(12):1131-41. doi: 10.1056/NEJMoa1607887. Epub 2016 Aug 30. PMID 27573206
- [Result] Birocchi S, Fiorelli EM, Podda GM. Andexanet Alfa for Factor Xa Inhibitor Reversal. N Engl J Med. 2016 Dec 22;375(25):2498-9. doi: 10.1056/NEJMc1613270. No abstract available. PMID 28009495
- [Result] Connolly SJ, Crowther M, Eikelboom JW, Gibson CM, Curnutte JT, Lawrence JH, Yue P, Bronson MD, Lu G, Conley PB, Verhamme P, Schmidt J, Middeldorp S, Cohen AT, Beyer-Westendorf J, Albaladejo P, Lopez-Sendon J, Demchuk AM, Pallin DJ, Concha M, Goodman S, Leeds J, Souza S, Siegal DM, Zotova E, Meeks B, Ahmad S, Nakamya J, Milling TJ Jr; ANNEXA-4 Investigators. Full Study Report of Andexanet Alfa for Bleeding Associated with Factor Xa Inhibitors. N Engl J Med. 2019 Apr 4;380(14):1326-1335. doi: 10.1056/NEJMoa1814051. Epub 2019 Feb 7. PMID 30730782
- [Derived] Milling TJ Jr, Middeldorp S, Xu L, Koch B, Demchuk A, Eikelboom JW, Verhamme P, Cohen AT, Beyer-Westendorf J, Gibson CM, Lopez-Sendon J, Crowther M, Shoamanesh A, Coppens M, Schmidt J, Albaladejo P, Connolly SJ; ANNEXA-4 Investigators. Final Study Report of Andexanet Alfa for Major Bleeding With Factor Xa Inhibitors. Circulation. 2023 Mar 28;147(13):1026-1038. doi: 10.1161/CIRCULATIONAHA.121.057844. Epub 2023 Feb 20. PMID 36802876
- [Derived] Costa OS, Connolly SJ, Sharma M, Beyer-Westendorf J, Christoph MJ, Lovelace B, Coleman CI. Andexanet alfa versus four-factor prothrombin complex concentrate for the reversal of apixaban- or rivaroxaban-associated intracranial hemorrhage: a propensity score-overlap weighted analysis. Crit Care. 2022 Jun 16;26(1):180. doi: 10.1186/s13054-022-04043-8. PMID 35710578
- [Derived] Huttner HB, Gerner ST, Kuramatsu JB, Connolly SJ, Beyer-Westendorf J, Demchuk AM, Middeldorp S, Zotova E, Altevers J, Andersohn F, Christoph MJ, Yue P, Stross L, Schwab S. Hematoma Expansion and Clinical Outcomes in Patients With Factor-Xa Inhibitor-Related Atraumatic Intracerebral Hemorrhage Treated Within the ANNEXA-4 Trial Versus Real-World Usual Care. Stroke. 2022 Feb;53(2):532-543. doi: 10.1161/STROKEAHA.121.034572. Epub 2021 Oct 14. PMID 34645283
- [Derived] Demchuk AM, Yue P, Zotova E, Nakamya J, Xu L, Milling TJ Jr, Ohara T, Goldstein JN, Middeldorp S, Verhamme P, Lopez-Sendon JL, Conley PB, Curnutte JT, Eikelboom JW, Crowther M, Connolly SJ; ANNEXA-4 Investigators. Hemostatic Efficacy and Anti-FXa (Factor Xa) Reversal With Andexanet Alfa in Intracranial Hemorrhage: ANNEXA-4 Substudy. Stroke. 2021 Jun;52(6):2096-2105. doi: 10.1161/STROKEAHA.120.030565. Epub 2021 May 10. PMID 33966491
- See also: Neurocrit Care. 2019;31:S37 — https://doi.org/10.1007/s12028-019-00857-7
- See also: Neurocrit Care. 2019;31:S222 — https://doi.org/10.1007/s12028-019-00857-7

RESULTS

PARTICIPANT FLOW:
Groups:
- Andexanet: Participants received andexanet as an intravenous (IV) bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- Andexanet - Additional Participants: Two additional participants received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes. Data from these 2 participants were obtained and evaluated after the data cutoff date of 30-June-2020 and, as such, are presented separately.
Period: Overall Study
Arm/Group | Andexanet | Andexanet - Additional Participants
Started | 477 | 2
Received At Least 1 Dose of Study Drug (Safety Population) | 477 | 2
Efficacy Population (All participants who received at least 1 dose of study drug and who met protocol-specified criteria for bleeding and anti-factor Xa (fXa) levels.) | 347 | 2
Death (These deaths occurred during the follow-up period.) | 3 | 0
Completed | 392 | 2
Not Completed | 85 | 0
Not completed — Death | 78 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received any amount of andexanet.
Groups:
- Total: Total of all reporting groups
Arm/Group | Andexanet | Andexanet - Additional Participants | Total
Number analyzed (Participants) | 477 | 2 | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (10.66) | 71.0 (11.31) | 77.9 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 1 | 219
  Male | 259 | 1 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 0 | 16
  Not Hispanic or Latino | 449 | 2 | 451
  Unknown or Not Reported | 12 | 0 | 12
Race/Ethnicity, Customized [Number; unit: participants] — Asian participants and American Indian or Alaska Native participants are reported as Other.
  participants
    Race : White | 414 | 0 | 414
    Race : Black or African American | 29 | 0 | 29
    Race : Other | 25 | 2 | 27
    Race : Missing | 9 | 0 | 9
Region of Enrollment [Number; unit: participants]
  North America | 212 | 0 | 212
  Europe | 248 | 0 | 248
  Japan | 17 | 2 | 19
FXa Inhibitor [Count of Participants; unit: Participants]
  Apixaban | 245 | 0 | 245
  Rivaroxaban | 174 | 2 | 176
  Edoxaban | 36 | 0 | 36
  Enoxaparin | 22 | 0 | 22
Bleed Type [Count of Participants; unit: Participants] — Endpoint Adjudication Committee (EAC) determined if each participant met the bleeding entry criteria for inclusion in the Efficacy Population.
  Participants
    Gastrointestinal | 109 | 0 | 109
    Intracranial Hemorrhage | 329 | 2 | 331
    Other | 39 | 0 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline In Anti-fXa Activity By FXa Inhibitor
Description: Anti-fXa activity was measured to assess the ability of andexanet to reverse the anticoagulant effect of FXa inhibitors. Baseline was defined as the last value obtained prior to the start of the andexanet bolus. The change from baseline was calculated as the reduction in anti-fXa activity from baseline to the on-treatment nadir (that is, the minimum value between end of bolus and end of infusion). Percent reduction was calculated as the ratio between the maximum change from baseline and the baseline value, multiplied by 100.
Time Frame: Baseline, 12 Hours (post infusion)
Population: Efficacy Population: all participants who received any amount of andexanet, met clinical bleeding criteria, and had an anti-fXa level of ≥75 nanograms/milliliter (ng/mL) for apixaban and rivaroxaban, ≥40 ng/mL for edoxaban, and ≥0.25 international units (IU)/mL for enoxaparin.
Measure: Median (95% Confidence Interval); unit: Percent Change
Groups:
- FXa Inhibitor: Apixaban: Participants who had recently received FXa inhibitor apixaban received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- FXa Inhibitor: Rivaroxaban: Participants who had recently received FXa inhibitor rivaroxaban received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- FXa Inhibitor: Edoxaban: Participants who had recently received FXa inhibitor edoxaban received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- FXa Inhibitor: Enoxaparin: Participants who had recently received FXa inhibitor enoxaparin received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- FXa Inhibitor: Rivaroxaban - Additional Participants: Two additional participants who had recently received FXa inhibitor rivaroxaban received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes. Data from these 2 participants were obtained and evaluated after the data cutoff date of 30-June-2020 and, as such, are presented separately.
Arm/Group | FXa Inhibitor: Apixaban | FXa Inhibitor: Rivaroxaban | FXa Inhibitor: Edoxaban | FXa Inhibitor: Enoxaparin | FXa Inhibitor: Rivaroxaban - Additional Participants
Number analyzed (Participants) | 169 | 130 | 28 | 17 | 2
Percent Change | -93.3 [-94.2 to -92.5] | -94.1 [-95.1 to -93.0] | -71.3 [-82.3 to -65.2] | -75.41 [-79.17 to -66.67] | -96.3 [-98.3 to -94.3]

2. Primary Outcome: Participants Achieving Hemostatic Efficacy
Description: Hemostatic efficacy was achieved when the body had time to produce thrombin and a subsequent clot and was rated by the EAC as: excellent; good; poor/none; not evaluable due to non-administrative reasons; not evaluable due to administrative reasons. These ratings were based on pre-specified criteria that were included in the EAC Charter. The EAC was blinded to anti-fXa activity levels. Participant results were classified as either success or failure based on the hemostatic efficacy rating (success = excellent/good, failure = poor/none). Participants rated by the EAC as non-evaluable due to administrative reasons were excluded from the analysis of hemostatic efficacy.
Time Frame: 12 Hours (post infusion)
Population: Efficacy Population: all participants who received any amount of andexanet, met clinical bleeding criteria, and had an anti-fXa level of ≥75 ng/mL for apixaban and rivaroxaban, ≥40 ng/mL for edoxaban, and ≥0.25 IU/mL for enoxaparin.
Measure: Count of Participants; unit: Participants
Groups:
- Bleed Type: Gastrointestinal: Participants with gastrointestinal bleeding who had recently received an FXa inhibitor received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- Bleed Type: Intracranial Hemorrhage: Participants with an intracranial hemorrhage who had recently received an FXa inhibitor received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- Bleed Type: Other: Participants with other types of bleeding who had recently received an FXa inhibitor received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes.
- Andexanet: Low Dose: Participants who had recently received FXa inhibitors received andexanet as an IV 400-mg bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion of 480 mg (4 mg/minute) administered over ~120 minutes.
- Andexanet: High Dose: Participants who had recently received FXa inhibitors received andexanet as an IV 800-mg bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion of 960 mg (8 mg/minute) administered over ~120 minutes.
- Overall: Participants who had recently received FXa inhibitor received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes. Does not include the 2 additional participants whose data were obtained and evaluated after the data cutoff date of 30-June-2020.
- Bleed Type: Intracranial Hemorrhage - Additional Participants: Two additional participants with an intracranial hemorrhage who had recently received an FXa inhibitor received andexanet as an IV bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion administered over ~120 minutes. Data from these 2 participants were obtained and evaluated after the data cutoff date of 30-June-2020 and, as such, are presented separately.
- Andexanet: Low Dose - Additional Participant: One additional participant who had recently received FXa inhibitors received andexanet as an IV 400-mg bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion of 480 mg (4 mg/minute) administered over ~120 minutes. Data from this participant were obtained and evaluated after the data cutoff date of 30-June-2020 and, as such, are presented separately.
- Andexanet: High Dose - Additional Participant: One additional participant who had recently received FXa inhibitors received andexanet as an IV 800-mg bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion of 960 mg (8 mg/minute) administered over ~120 minutes. Data from this participant were obtained and evaluated after the data cutoff date of 30-June-2020 and, as such, are presented separately.
Arm/Group | FXa Inhibitor: Apixaban | FXa Inhibitor: Rivaroxaban | FXa Inhibitor: Edoxaban | FXa Inhibitor: Enoxaparin | Bleed Type: Gastrointestinal | Bleed Type: Intracranial Hemorrhage | Bleed Type: Other | Andexanet: Low Dose | Andexanet: High Dose | Overall | FXa Inhibitor: Rivaroxaban - Additional Participants | Bleed Type: Intracranial Hemorrhage - Additional Participants | Andexanet: Low Dose - Additional Participant | Andexanet: High Dose - Additional Participant
Number analyzed (Participants) | 169 | 127 | 28 | 16 | 74 | 244 | 22 | 269 | 71 | 340 | 2 | 2 | 1 | 1
Participants
  Excellent/Good | 134 | 102 | 22 | 14 | 61 | 193 | 18 | 218 | 54 | 272 | 2 | 2 | 1 | 1
  Poor/None | 35 | 25 | 6 | 2 | 13 | 51 | 4 | 51 | 17 | 68 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percent Change From Baseline In Anti-fXa Activity By Hemostatic Efficacy
Description: This outcome measure assessed the relationship between hemostatic efficacy and anti-fXa activity in participants receiving an FXa inhibitor who had acute major bleeding. Anti-fXa activity was measured to assess the ability of andexanet to reverse the anticoagulant effect of FXa inhibitors. Baseline was defined as the last value obtained prior to the start of the andexanet bolus. Hemostatic efficacy was achieved when the body had time to produce thrombin and a subsequent clot and was rated by the EAC as: excellent; good; poor/none; not evaluable due to non-administrative reasons; not evaluable due to administrative reasons.
Time Frame: Baseline, 12 Hours (post infusion)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | FXa Inhibitor: Apixaban | FXa Inhibitor: Rivaroxaban | FXa Inhibitor: Edoxaban | FXa Inhibitor: Enoxaparin | FXa Inhibitor: Rivaroxaban - Additional Participants
Number analyzed (Participants) | 169 | 127 | 28 | 16 | 2
Percent Change
  Excellent/Good: number analyzed (Participants) | 134 | 102 | 22 | 14 | 2
  Excellent/Good | -93.4 [-94.3 to -92.6] | -94.6 [-95.2 to -93.5] | -75.8 [-84.4 to -65.2] | -75.20 [-77.08 to -65.91] | -96.3 [-98.3 to -94.3]
  Poor/None: number analyzed (Participants) | 35 | 25 | 6 | 2 | 0
  Poor/None | -93.3 [-95.3 to -90.6] | -92.4 [-96.5 to -85.0] | -65.2 [-85.3 to 3.0] | -78.44 [-82.46 to -74.42] |

ADVERSE EVENTS:
Time Frame: Day 1 through Day 37.
Groups:
- Andexanet: High Dose: Participants who had recently received FXa inhibitors received andexanet as an IV 800- mg bolus administered over ~15 to 30 minutes, followed immediately by a continuous infusion of 960 mg (8 mg/minute) administered over ~120 minutes.
Arm/Group | Andexanet: Low Dose | Andexanet: High Dose
All-Cause Mortality (participants affected / at risk) | 66/382 | 15/97
Serious Adverse Events (participants affected / at risk) | 157/382 | 43/97
Other Adverse Events (participants affected / at risk) | 40/382 | 8/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Andexanet: Low Dose (N=382) | Andexanet: High Dose (N=97)
Ischaemic Stroke (Nervous system disorders) | 8 (8) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 4 (4) | 4 (4)
Haemorrhage Intracranial (Nervous system disorders) | 7 (7) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 5 (5) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 4 (4) | 1 (1)
Neurological Decompensation (Nervous system disorders) | 2 (2) | 2 (2)
Intraventricular Haemorrhage (Nervous system disorders) | 3 (3) | 0/2 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 2 (2) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial Venous Sinus Thrombosis (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Altered State Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Basal Ganglia Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basilar Artery Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Brain Compression (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar Ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Ventricle Dilatation (Nervous system disorders) | 0 (0) | 1 (1)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0/2 (0)
Facial Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal Nerve Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Slow Response To Stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (15) | 6 (6)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Septic Shock (Infections and infestations) | 4 (4) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
CNS Ventriculitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Serratia Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subdural Empyema (Infections and infestations) | 1 (1) | 0 (0)
Tracheostomy Infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 3 (3) | 3 (3)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 4 (4) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 5 (6) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Aorto-Duodenal Fistula (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Iliac Artery Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 3 (3) | 2 (2)
General Physical Health Deterioration (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Brain Herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaplastic Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CSF Red Blood Cell Count Positive (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0)
Electroencephalogram Abnormal (Investigations) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
Troponin I Increased (Investigations) | 0 (0) | 1 (1)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 2 (2) | 0 (0)
Mental Disorder Due To A General Medical Condition (Psychiatric disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Social Stay Hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Ventricular Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Andexanet: Low Dose (N=382) | Andexanet: High Dose (N=97)
Urinary Tract Infection (Infections and infestations) | 40 (40) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT02329327/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT02329327/SAP_001.pdf